CLINICAL TRIAL: NCT06248281
Title: Be Cool: An Innovative and Holistic Psychoeducational Program to Improve and Promote Care, Education and Quality of Life for Multiple Sclerosis Individuals
Brief Title: Be Cool: An Innovative and Holistic Psychoeducational Program for Multiple Sclerosis Individuals
Acronym: BeCool
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: Greek Multiple Sclerosis Society (Unknown); European Committee for Treatment and Research in Multiple Sclerosis (Unknown)
Responsible Party: Principal Investigator, Antonia Kaltsatou, PhD, Adjunct Lecturer, University of Thessaly
Other Study IDs: 396/23
Record Dates: First submitted 2023-12-18; First posted 2024-02-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: symptom management; hybrid program; rehabilitation; quality of life; psychoeducational program
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cryotherapy; Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: The experimental group will attend a structured psychoeducational program developed to build and promote psychological flexibility. In combination with this, participants of this group will have to follow a head and neck cooling protocol. Also, participants of this group will be required to increase their habitual exercise levels and follow a video exercise program specifically designed for their needs and improve their nutrition based on the instructions of a nutritionist and videos specially designed for them.
  Interventions: Other: combination of different rehabilitation strategies
- Control group: As per the study plan, the Control group has been designated as the control group. They will continue with their normal lifestyle without any participation in rehabilitation activities or programs.
  Interventions: Other: combination of different rehabilitation strategies

INTERVENTIONS:
Other: combination of different rehabilitation strategies — The psychoeducational program will be conducted through weekly online video-conferencing group sessions that will last for two hours. In addition to these sessions, participants will receive psychoeducational material such as readings, videos, podcasts, worksheets, and homework exercises every week. This material will allow participants to practice at their own pace during the session intervals.
  The exercise training program for individuals with MS will be tailored to meet the unique and individual needs of each participant. To achieve this, a head and neck cooling protocol will be implemented using commercially available cooling equipment, specifically the Headcool Power and Neckcool Tie from Inuteq. Participants will need to wear the cooling cup and neck wrap for two hours daily. The equipment will be activated using 10°C tap water. Finally, a nutritionist will provide personalized nutritional guidance including weekly diet observation and recipe videos.
  Other Names: cooling therapy; diet; phycology-behavioral-mindfulness intervention; exercise traiining

SUMMARY:
This observational study aims to investigate the impact of an online psychoeducational program, combined with cooling therapy, nutrition, psychological intervention, and exercise, on the resilience, treatment adherence, symptom management, and quality of life of individuals with Multiple Sclerosis. The study will last for six months, during which two groups of 15 participants with similar characteristics and a diagnosis of Multiple Sclerosis will take part in the protocol. Group A will follow the research protocol, while Group B, the Control group, will not participate in any rehabilitation intervention.

DETAILED DESCRIPTION:
Fifteen individuals with multiple sclerosis will participate in an innovative, hybrid rehabilitation program, encompassing several key components to enhance their well-being. The program includes:

1. Exercise Intervention: Participants will engage in specially designed exercise programs. Every two weeks, they will meet virtually with an exercise physiologist via Microsoft Teams for tailored education about their specific needs. Additionally, a customized exercise video will be uploaded weekly to the Teams platform, ensuring ongoing physical engagement.
2. Nutritional Evaluation and Education: Nutrition is a core focus. A nutritionist will meet with the participants bi-weekly to discuss their dietary needs and educate them on maintaining a balanced diet to support their condition. Further enhancing this aspect, a nutritious recipe will be uploaded to the platform each week, offering practical dietary guidance.
3. Psychological Support: Psychological well-being is addressed through weekly group meetings conducted by a psychologist. These sessions will utilize Acceptance and Commitment Therapy (ACT) strategies to help participants manage their symptoms, accept their condition, and improve their overall quality of life.
4. Head and Neck Cooling Strategy: Recognizing the importance of temperature regulation in MS, participants will be advised to apply a cooling strategy to the head and neck area for at least two hours daily, providing symptomatic relief.

To monitor progress and adjust the program as needed, participants' functional ability, nutritional status, psychological condition, and overall quality of life will be evaluated at three key points: baseline (before starting the program), at the three-month mark, and upon completion of the program at six months.

This program is structured to provide a holistic, supportive, and adaptable approach to managing multiple sclerosis, focusing on physical health, nutritional balance, psychological support, and practical strategies for daily living.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have been diagnosed with MS using the McDonald criteria, ensuring a standardized and validated diagnostic approach.
2. Participants should have been relapse-free during the six months leading up to the study to avoid potential confounding factors.
3. Participants must have no musculoskeletal impediment that could affect their ability to engage in the exercise component of the program.
4. Participants must have a score on the Expanded Disability Status Scale (EDSS) ranging from 0 to 5.5, indicating ambulatory ability without the need for a cane for at least 100 meters.
5. Participants should have a history of sensitivity to heat, as reported by their treating physician, justifying the need for cooling therapy as part of the hybrid program.
6. Participants must not have used cooling therapy or participated in any form of exercise training for at least four months prior to their participation in the study.

   -

Exclusion Criteria:

1. Previously diagnosed conditions known to impact physiological responses to heat exposure, including diabetes mellitus, hypertension, heart disease, or kidney disease.
2. Use of medications to manage MS-related symptoms, such as antidepressants, psychostimulants, anticonvulsants, antispasmodics, and anticholinergic drugs.

   -

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the GMSS (https://gmss.gr/) based on specific inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
anxiety and depression | Baseline, after three months and at the end of the six months
  This will be estimated with the "The Hospital Anxiety and Depression Scale - HADS". The Hospital Anxiety and Depression Scale (HADS) is a widely used questionnaire specifically designed to identify and measure the levels of anxiety and depression in individuals. It is particularly useful in medical settings, as it helps distinguish between psychological distress and physical illness.
Overall quality of life, namely satisfaction with their life | Baseline, after three months and at the end of the six months
  This will be estimated with the questionnaire of Multiple Sclerosis Quality of Life-54 (MSQOL-54)
Perception of stress | Baseline, after three months and at the end of the six months
  Perceived Stress Scale (PSS) will be used. This is a widely used psychological instrument for measuring the perception of stress. It assesses the degree to which situations in one's life are appraised as stressful. Items on the PSS ask about feelings and thoughts during the last month, and scores on the PSS can range from 0 to 40, with higher scores indicating higher perceived stress.
Cognitive fusion which refers to the degree to which an individual's thoughts and feelings are intertwined with their sense of self, often leading to an inability to separate from, or 'defuse' from, these internal experiences. | Baseline, after three months and at the end of the six months
  The Cognitive Fusion Questionnaire (CFQ-7) questionnaire that measures cognitive fusion, which a key concept in Acceptance and Commitment Therapy (ACT) will be used. The CFQ-7, with its 7 items, assesses the extent to which a person experiences this phenomenon.
The value of living | Baseline, after three months and at the end of the six months
  The Valued Living Questionnaire (VLQ) will be used. The VLQ is designed to assess valued living, which is another core concept in ACT. It helps individuals to identify what is truly important and meaningful to them in various domains of life (such as family, career, health) and to what extent they have been living in accordance with these values.
Psychological flexibility which is the ability to be in the present moment with full awareness and openness to experiences, and to take action guided by one's values. | Baseline, after three months and at the end of the six months
  The MPFI-Psychological Flexibility Subscale will be used. This subscale is part of a larger questionnaire and specifically measures psychological flexibility, an essential aspect of mental health and well-being.
The resilience which is defined as the ability to cope with and bounce back from adversity. | Baseline, after three months and at the end of the six months
  The Connor-Davidson Resilience Scale (CDRISC-25) will be used. This 25-item scale measures resilience, defined as the ability to cope with and bounce back from adversity. Higher scores indicate greater resilience.
Aerobic capacity and ability to walk | Baseline, after three months and at the end of the six months
  The Two Minute Walk Test (2MWT) is a simple, easy-to-administer functional exercise test used primarily in clinical settings. It measures the distance an individual is able to walk on a flat, hard surface in a period of two minutes.
Lower body strength and functional mobility | Baseline, after three months and at the end of the six months
  The Five Times Sit to Stand Test (5xSST) will be used which is a simple yet effective physical performance test used primarily to assess lower body strength and functional mobility. The test involves timing how long it takes an individual to stand up and sit down five times as quickly as possible from a standard height chair without using their arms for support. A longer time to complete the test generally indicates lower functional performance.
Static and dynamic balance ability | Baseline, after three months and at the end of the six months
  The Berg Balance Scale (BBS) will be used which is a widely used clinical test of a person's static and dynamic balance abilities. It is particularly common in elderly populations and among those recovering from injury or dealing with conditions that affect balance.
Mobility and walking speed | Baseline, after three months and at the end of the six months
  The Timed 25-Foot Walk (T25-FW) will be used which is a functional test commonly used to assess mobility and walking speed in individuals, particularly those with neurological conditions such as multiple sclerosis (MS).The test involves timing how quickly a person can walk 25 feet at their usual pace, usually conducted along a flat, straight course.

SECONDARY OUTCOMES:
Finger dexterity and arm-hand coordination | Baseline, after three months and at the end of the six months
  The 9-Hole Peg Test (9-HPT) will be used which is a standardized, widely used assessment tool in clinical and research settings to measure finger dexterity and arm-hand coordination. It's particularly useful for evaluating upper extremity function in individuals with neurological conditions, such as multiple sclerosis (MS) and stroke.
Core temperature | Baseline, after three months and at the end of the six months
  With a gastrointestinal telemetric capsule (e-Celsius)
Skin temperature | Baseline, after three months and at the end of the six months
  iButtons
Nutritional status, how balance is their nutrition | Baseline, after three months and at the end of the six months
  This will be estimated with questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios Orologas, MD, PhD, Study Chair — Greek Multiple Sclerosis Society
Locations (1):
- Greek Multiple Sclerosis Society, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No
Once the protocol is completed and published, all the data will be available upon request to other researchers.

REFERENCES:
- [Background] Kaltsatou A, Flouris AD. Impact of pre-cooling therapy on the physical performance and functional capacity of multiple sclerosis patients: A systematic review. Mult Scler Relat Disord. 2019 Jan;27:419-423. doi: 10.1016/j.msard.2018.11.013. Epub 2018 Nov 13. PMID 30544086